CLINICAL TRIAL: NCT04379024
Title: Pilot Study of Effects of Duavee® on Imaging and Blood Biomarkers In Women With Menopausal Symptoms at Increased Risk for Breast Cancer
Brief Title: Pilot Study of Effects of Duavee® on Imaging and Blood Biomarkers In Women With Menopausal Symptoms
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study agent no longer available
Sponsor: Carol Fabian, MD (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study00145121
Record Dates: First submitted 2020-05-03; First posted 2020-05-07 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-03

CONDITIONS: Focus of Study is Healthy Women at Risk for Breast Cancer
Keywords: Imaging; Biomarkers
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Intervention Model Description: Randomized to active agent or wait-list control.
Masking Description: Randomization assignment is masked to all roles prior to randomization. Subsequent to randomization, agent is dispensed open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate active agent (Experimental): Duavee. One capsule daily for 6 months (+/- 1 month) of Duavee (Bazedoxifene 20 mg plus conjugated estrogens 0.45 mg)
  Interventions: Drug: DUAVEE 0.45Mg-20Mg Tablet
- Delayed active agent (Other): No intervention for first 6 months. Then option to receive daily Duavee for 6 months.
  Interventions: Drug: DUAVEE 0.45Mg-20Mg Tablet

INTERVENTIONS:
Drug: DUAVEE 0.45Mg-20Mg Tablet — One capsule daily for 6 months (+/- 1 month)
  Other Names: Bazedoxifene 20 mg plus conjugated estrogens 0.45 mg

SUMMARY:
Pilot study to test feasibility of 6 months of Duavee® vs wait-list control in post-menopausal women symptomatic for hot flashes.

DETAILED DESCRIPTION:
Duavee® which is the combination of the selective estrogen receptor modulator bazedoxifene and conjugated estrogen 0.45 mg) is an FDA approved drug for treatment of hot-flashes and prevention of osteoporosis in postmenopausal women. The investigators recently reported the results of a single arm pilot study suggesting that 6 months of Duavee® was associated with improvement in several risk biomarkers including benign breast tissue proliferation, mammographic fibroglandular volume, IGF-1, SHBG and progesterone in high risk women in late menopause transition. Prior to opening a randomized Phase IIB trial of 6 months of Duavee® vs placebo in high risk women with hot-flashes followed by open label Duavee®, the intent of this study is to assess probable uptake of such a trial design with a pilot of 6 months of Duavee® vs wait-list control in symptomatic women. Additional imaging biomarker information from MRI will be obtained. A finding on MRI of greater background parenchymal enhancement (BPE) in high risk women is positively associated with higher probability of developing breast cancer and is independent of fibroglandular volume. BPE is reduced by selective estrogen receptor modulators including tamoxifen. The investigators will investigate change in MRI BPE over time for women randomly assigned to either receive Duavee® or not (wait-list control). The investigators will also explore development of fully automated breast MRI volumetric density measures.

ELIGIBILITY:
Inclusion Criteria:

* Women who report vasomotor symptoms (hot flashes or night sweats)
* No menstrual periods for at least 3 months
* Must have at least one ovary (hysterectomy is permitted; bilateral salpingo- oophorectomy is excluded).
* BMI <36 kg/m2
* Moderate risk of developing breast cancer based on having any one or more of the following:

  * First or 2nd degree relative with breast cancer
  * Known carrier of moderate to high penetrance germline mutation
  * Prior breast biopsy showing proliferative breast disease or multiple biopsies
  * High mammographic density (Volpara® categories c or d or BIRADs density assessment as heterogeneously or extremely dense (c or d).
  * IBIS Breast Cancer Risk Evaluation Version 8 10-year relative risk of >2X that for the population for age group.

Exclusion Criteria:

* Risk: A prior biopsy showing LCIS, DCIS, or invasive breast cancer.
* Medical Conditions:

  * Have a predisposition to or prior history of thromboembolism, deep venous thrombosis, pulmonary embolism, or stroke
  * History of renal or liver disease
  * Prior invasive ovarian or endometrial cancer
* Medications

  * Current anticoagulant use other than low dose aspirin
  * Taking systemic hormones within two months (eight weeks) prior to baseline MRI and mammogram.
  * Taking tamoxifen, raloxifene, Duavee, or any selective estrogen receptor modulator, or an aromatase inhibitor within 12 months prior to baseline MRI and mammogram.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Number of potential participants who consent to enrollment | Enrollment
  Trial design is acceptable to potential subjects, as evidenced by participation

SECONDARY OUTCOMES:
Change in breast background parenchymal enhancement (BPE) | 6 months
  BPE assessed by abbreviated MRI at baseline and after 6 months
Change in fibroglandular volume (FGV) | 6 months
  FGV assessed by Volpara software on 3D mammograms acquired at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabian CJ, Nye L, Powers KR, Nydegger JL, Kreutzjans AL, Phillips TA, Metheny T, Winblad O, Zalles CM, Hagan CR, Goodman ML, Gajewski BJ, Koestler DC, Chalise P, Kimler BF. Effect of Bazedoxifene and Conjugated Estrogen (Duavee) on Breast Cancer Risk Biomarkers in High-Risk Women: A Pilot Study. Cancer Prev Res (Phila). 2019 Oct;12(10):711-720. doi: 10.1158/1940-6207.CAPR-19-0315. Epub 2019 Aug 16. PMID 31420361